CLINICAL TRIAL: NCT05768360
Title: A Phase I, Fixed-sequence, Open-label Study to Assess the Effects of Savolitinib on the Pharmacokinetics of Substrates of Human Transporters Digoxin (P-gp), Rosuvastatin (OATP1B1/3), Metformin (OCT2, MATE1/2K), and Furosemide (OAT1/3) in Healthy Male Subjects
Brief Title: A Study to Assess the Effects of Savolitinib on the Pharmacokinetics of Digoxin, Rosuvastatin, Metformin, and Furosemide in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: D5084C00014; 2022-003785-21 (EudraCT Number)
Record Dates: First submitted 2023-03-03; First posted 2023-03-14 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Healthy Male Subjects
Keywords: Drug-Drug Interaction; Substrate of human drug transporters; Fixed-sequence; Drug cocktail
MeSH Terms: interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Digoxin; Metformin; Rosuvastatin Calcium; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug cocktail/Savolitinib + Drug cocktail (Experimental): Subjects will receive two different interventions in two periods (Periods 1 and 2). In Period 1, the subjects will receive a single-dose of Drug cocktail components (digoxin Dose B, furosemide Dose C, metformin hydrochloride Dose D, and rosuvastatin Dose E). During Period 2, the subjects will receive savolitinib dose A in combination with the Drug cocktail components.
  Interventions: Drug: Savolitinib; Drug: Digoxin; Drug: Metformin Hydrochloride; Drug: Rosuvastatin; Drug: Furosemide

INTERVENTIONS:
Drug: Savolitinib — The subjects will receive single dose of oral film-coated tablet of Savolitinib A dose on Day 1 of Period 2 within 25 minutes [+ 5 minutes] from the start of meal.
Drug: Digoxin — The subjects will receive single dose of oral uncoated tablet of Digoxin Dose B on Day 1 of Period 1 and Period 2 within 25 minutes [+ 5 minutes] from the start of meal.
Drug: Metformin Hydrochloride — The subjects will receive single dose of oral film-coated tablet of Metformin Hydrochloride Dose D on Day 1 of Period 1 and Period 2 within 25 minutes [+ 5 minutes] from the start of meal.
Drug: Rosuvastatin — The subjects will receive single dose of oral film-coated tablet of Rosuvastatin Dose E on Day 1 of Period 1 and Period 2 within 25 minutes [+ 5 minutes] from the start of meal.
Drug: Furosemide — The subjects will receive single dose of oral solution of Furosemide Dose C on Day 1 of Period 1 and Period 2 within 25 minutes [+ 5 minutes] from the start of meal.

SUMMARY:
This study will assess the effects of savolitinib on the pharmacokinetics (PK) of substrates of human transporters digoxin (P-gp), rosuvastatin (OATP1B1/3), metformin (OCT2, MATE1/2K), and furosemide (OAT1/3) in healthy male subjects, performed at a single clinical unit.

DETAILED DESCRIPTION:
This study will be performed at a single clinical unit.

Subjects will be admitted to the clinical unit on Day -1 of Period 1 and Period 2. Subjects will have a washout period of 14 days between Period 1 and Period 2.

Period 1: Subjects will recieve a single dose of a drug cocktail of 4 medications (digoxin Dose B, furosemide Dose C, metformin hydrochloride Dose D, and rosuvastatin Dose E).

Period 2: Participants will receive savolitinib (Dose A) in combination with the drug cocktail of 4 medications as received in Period 1.

The study will consist of 4 visits:

Visit 1 (Enrollment): Following full written informed consent, subjects will be screened for eligibility.

Visit 2 (Period 1: Treatment and Sample Collection Period): Each subject will be admitted to the clinical unit on Day -1 of Period 1, single dose of drug cocktail is administered on Day 1, and remain in clinical unit until Day 5 assessments. A washout period of 14 days is followed.

Visit 3 (Period 2: Treatment and Sample Collection Period): Each subject will be admitted to the clinical unit on Day -1 of Period 2, single dose of savolitinib and drug cocktail is administered, and remain in clinical unit until Day 5 assessments.

Visit 4 (Follow-up): Subjects will attend the clinical unit for a final Follow-up Visit 5 to 7 days post Day 5 in Period 2.

Each subject will be involved in the study for 9 weeks including screening to final follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects must use barrier contraception (condoms) during sexual intercourse with a female partner of childbearing potential during the study and for 6 months after the last dose of the IMPs investigational medical products (IMPs).
2. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
3. Regular bowel movements (ie, on average production of at least 1 stool per day).

Exclusion Criteria:

1. History of any clinically significant disease or disorder
2. History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results.
4. Any clinically significant abnormalities on 12-lead electrocardiogram (ECG) at screening and/or first admission to the clinical unit, as judged by the investigator.
5. QTcF >450 ms or QT ≥500 ms or other ECG abnormality making interpretation more difficult, as judged by the investigator, or a history of additional risk factors for Torsades de Points (eg heart failure, hypokalemia, family history of long QT syndrome), which in the opinion of the investigator may put the subject at risk.
6. Any positive result on screening for serum hepatitis B surface antigen OR anti-HBc antibody, indicative of active hepatitis B (ie, subjects with positive anti-HBc antibody result are acceptable if anti HBc IgM antibodies are negative), hepatitis C antibody, and HIV antibody.
7. History of latent or chronic infections (eg, tuberculosis, recurrent sinusitis, genital herpes, urinary tract infections) or at risk of infection.
8. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months (12 weeks) or within 5 half-lives of the drug, whichever is longer, of Visit 2 (Day -1 of Period 1) in this study or participation in a method development study (no drug) 1 month prior to Visit 2. The period of exclusion ends 3 months after the final dose or after 5 elimination half-lives of the drug or 1 month after the last visit, whichever is the longer.
9. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to savolitinib, or drug cocktail medications or their excipients.
10. Subject has clinical signs and symptoms consistent with Coronavirus disease (COVID-19), eg, fever, dry cough, dyspnea, sore throat, fatigue, or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission unless confirmed by a negative severe acute respiratory syndrome coronavirus 2 polymerase chain reaction test (SARS-CoV-2 PCR test).
11. Vulnerable subjects, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
12. Positive screen for drugs of abuse or cotinine at screening or on each admission to the clinical unit or positive screen for alcohol on each admission to the clinical unit.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-06-24 (Actual)

PRIMARY OUTCOMES:
Plasma Area Under Concentration-time Curve from zero to infinity (AUCinf) of the drug cocktail components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To evaluate AUCinf of drug cocktail components when administered alone (period 1) and in combination with savolitinib (period 2)
Plasma Area under the concentration-curve from zero to the last quantifiable concentration (AUClast) of the drug cocktail components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To evaluate AUClast of drug cocktail components when administered alone (period 1) and in combination with savolitinib (period 2)
Plasma partial area under the concentration-time curve from time 0 to time t post-dose (AUC(0-t)) of the drug cocktail components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To evaluate (AUC(0-t)) of drug cocktail components when administered alone (period 1) and in combination with savolitinib (period 2).
Maximum observed plasma drug concentration (Cmax) of drug cocktail components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To evaluate Cmax of drug cocktail components when administered alone (period 1) and in combination with savolitinib (period 2).
The ratio of plasma AUCinf (R AUCinf) of the drug cocktail components in the presence and absence of savolitinib | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To evaluate AUCinf ratio of drug cocktail components when administered alone (period 1) and in combination with savolitinib (period 2).
The ratio of plasma AUC(0-t) (R AUC(0-t)) of the drug cocktail components in the presence and absence of savolitinib | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To evaluate AUC(0-t) ratio of drug cocktail components when administered alone (period 1) and in combination with savolitinib (period 2).
The ratio of plasma Cmax (R Cmax) of drug cocktail components in the presence and absence of savolitinib | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To evaluate Cmax ratio of drug cocktail components when administered alone (period 1) and in combination with savolitinib (period 2).

SECONDARY OUTCOMES:
Number of participants with adverse events | Day 1 in Periods 1 (Week 1) and 2 (Week 4) to Day 7 (follow-up after last Pharmacokinetic (PK) sample)
  To assess safety and tolerability of savolitinib following oral dosing.
Area under plasma concentration-time curve from zero to infinity (AUCinf) of savolitinib and its metabolites (M2 and M3) | Day 1 and Day 2 in Period 2 (Week 4)
  To assess AUCinf of savolitinib and its metabolites (M2 and M3).
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUCinflast) of savolitinib and its metabolites (M2 and M3) | Day 1 and Day 2 in Period 2 (Week 4)
  To assess AUClast of savolitinib and its metabolites (M2 and M3)
Partial area under the concentration-time curve from time 0 to time t post-dose (AUC(0-t)) of savolitinib and its metabolites (M2 and M3) | Day 1 and Day 2 in Period 2 (Week 4)
  To assess AUC(0-t) of savolitinib and its metabolites (M2 and M3).
Maximum observed plasma (peak) drug concentration (Cmax) of savolitinib and its metabolites (M2 and M3) of savolitinib and its metabolites (M2 and M3) | Day 1 and Day 2 in Period 2 (Week 4)
  To assess Cmax of savolitinib and its metabolites (M2 and M3).
Observed lowest concentration before the next dose is administered (Ctrough) of savolitinib and its metabolites (M2 and M3) | Day 1 and Day 2 in Period 2 (Week 4)
  To assess Ctrough of savolitinib and its metabolites (M2 and M3).
Terminal elimination half-life (t½λz) of savolitinib and its metabolites (M2 and M3) | Day 1 and Day 2 in Period 2 (Week 4)
  To assess t½λz of savolitinib and its metabolites (M2 and M3).
Time to reach maximum observed concentration (tmax) of savolitinib and its metabolites (M2 and M3) | Day 1 and Day 2 in Period 2 (Week 4)
  To assess tmax of savolitinib and its metabolites (M2 and M3).
Apparent volume of distribution based on the terminal phase (Vz/F) of savolitinib and its metabolites (M2 and M3) | Day 1 and Day 2 in Period 2 (Week 4)
  To assess Vz/F of savolitinib and its metabolites (M2 and M3).
Apparent total body clearance (CL/F) of savolitinib and its metabolites (M2 and M3) | Day 1 and Day 2 in Period 2 (Week 4)
  To assess CL/F of savolitinib and its metabolites (M2 and M3).
Maximum observed plasma (peak) drug concentration (Cmax) of cocktail parent components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To assess the Cmax of the drug cocktail parent components.
Time to reach maximum observed plasma concentration (Tmax) of the cocktail parent components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To assess the PK parameter tmax of the drug cocktail parent components
Plasma terminal elimination half-life (t½λz) of cocktail parent components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To assess the PK parameter t½λz of the drug cocktail parent components.
Plasma terminal rate constant, estimated by log-linear least squares regression of the terminal part of the concentration-time curve (λz) of cocktail parent components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To assess the PK parameter λz of the drug cocktail parent components.
Plasma Apparent total body clearance (CL/F) of cocktail parent components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To assess the PK parameter CL/F of the drug cocktail parent components.
Plasma Apparent volume of distribution based on the terminal phase (Vz/F) of cocktail parent components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To assess the PK parameter Vz/F of the drug cocktail parent components.
Renal clearance (CLR) of cocktail parent components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To assess the urine PK parameter CLR of the drug cocktail parent components.
Cumulative amount of unchanged drug excreted into urine (Ae) of cocktail parent components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To assess the urine PK parameter Ae of the drug cocktail parent components.
Cumulative amount of unchanged drug excreted into the urine from time 0 to time t (Ae(0-t)) of cocktail parent components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To assess Ae(0-t) of the drug cocktail parent components
Percentage of dose excreted unchanged in urine from time 0 to t (fe(0-t)) of cocktail parent components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To assess fe(0-t) of the drug cocktail parent components.
Cumulative amount of unchanged drug excreted into urine (CumAe) of the cocktail parent components | Day 1 to Day 5 in Periods 1 (Week 1) and 2 (Week 4)
  To assess CumAe of the drug cocktail parent components

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home